CLINICAL TRIAL: NCT06080789
Title: A Phase 2a, Multi-Center, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of a Single Dose of RABI-767 Administered by Endoscopic Ultrasound-Guided Peripancreatic Injection Plus Standard-of-Care Versus Standard-of-Care Only in Participants With Predicted Severe Acute Pancreatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of a Single Dose of RABI-767 in Participants With Acute Pancreatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Panafina, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RABI-767-201
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RABI-767 plus Standard-of-Care (Experimental): Single-dose 125 mg RABI-767 plus standard-of-care
  Interventions: Drug: RABI-767
- Standard-of-Care Only (No Intervention): No Intervention, Standard-of-Care Only

INTERVENTIONS:
Drug: RABI-767 — 125 mg single-dose given by endoscopic-ultrasound (EUS) guided peripancreatic injection.
  Arms: RABI-767 plus Standard-of-Care

SUMMARY:
The goal of this clinical trial is to test the safety and effectiveness of a single dose of RABI-767 given by endoscopic ultrasound (EUS) guided peripancreatic injection in participants with predicted severe acute pancreatitis.

The main question the study aims to answer is:

• Is a single-dose of RABI-767 given by EUS-guided peripancreatic injection safe in patients with predicted severe acute pancreatitis.

The study also aims to answer:

• Is a single-dose of RABI-767 given by EUS-guided peripancreatic injection effective in treating patients with predicted severe acute pancreatitis.

Study participants will be randomly assigned (like the flip of a coin) to receive a single dose of RABI-767 plus supportive care or supportive care only.

The study sponsor will compare safety and efficacy data collected from participants who receive RABI-767 to participants who receive supportive care only to test if RABI-767 is safe and effective.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of acute pancreatitis
* Predicted severe acute pancreatitis, based on protocol defined criteria
* Lack of clinically meaningful improvement from status at admission, at the discretion of Investigator, at the time of randomization
* Suitable for EUS-guided study drug administration procedure
* Contrast-enhanced computed tomography (CECT) or magnetic resonance imaging (MRI) of the abdomen/pancreas available for the evaluation of exclusion criteria

Key Exclusion Criteria:

* Confirmed severe acute pancreatitis as defined by the Revised Atlanta Classification of Acute Pancreatitis (ie, Persistent [> 48 hours] organ failure, per Modified Marshall Score), prior to randomization
* Anticipated discharge from hospital within 48 hours of randomization
* More than 30% pancreatic necrosis on screening CECT or MRI
* History of previous pancreatic necrosis, including necrosectomy
* History of calcific chronic pancreatitis
* Evidence of cholangitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Enrollment/Randomization to Day 28 (or hospital discharge, if earlier)
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the study intervention, regardless of its causal relationship to the study intervention. For the purposes of this study, any AE occurring in any study participant (regardless of treatment group assignment) at any time after enrollment/randomization, even if no study intervention has been administered, will be recorded.
Number of Participants with Serious Adverse Events | Enrollment/Randomization to Day 35 Follow-up
  A serious adverse event (SAE) is an AE, regardless of causality, that fulfills one or more protocol defined criteria for being serious.
Change from Baseline in Clinical Chemistry Parameters | Baseline to Day 7
Change from Baseline in Hematology Parameters | Baseline to Day 7
Change from Baseline in Vital Signs | Baseline to Day 7
Change from Baseline in Pulse Oximetry and Oxygen Delivery Measurements | Baseline to Day 7

SECONDARY OUTCOMES:
Development of Severe Acute Pancreatitis | Day 1 to Day 28 (or hospital discharge, if earlier)
  Defined as >48 hours persistent organ failure
Development of New Onset Moderately Severe Acute Pancreatitis | Day 1 to Day 28 (or hospital discharge, if earlier)
  Defined as transient organ failure and/or local or systemic complications without persistent organ failure
Development of Pancreatic Necrosis | Baseline to Day 60 Follow-up
  As identified on CECT/CEMRI imaging; may be further sub-grouped into <30%, 30%-50%, and >50% pancreatic necrosis, if data allow.
Development of Local Complications of Acute Pancreatitis | Baseline to Day 60 Follow-up
  As identified on CECT/CEMRI imaging; may be further sub-grouped by type of complication, if data allow.
Mortality due to acute pancreatitis and/or complications secondary to acute pancreatitis | Day 1 to Day 60 Follow-up
  Death caused by acute pancreatitis and/or complications secondary to acute pancreatitis
Mortality due to any cause | Day 1 to Day 60 Follow-up
  Death due to any cause
Days in Hospital | Day 1 through Day 28 (or hospital discharge, if earlier)
Re-hospitalization for acute pancreatitis or related complications | From initial hospital discharge to Day 35 Follow-up
  Number of participants re-hospitalized for acute pancreatitis or related complications out of total participants who are discharged.
Length of Stay in Intensive Care Unit | Day 1 through Day 28 (or hospital discharge, if earlier)
Development of New Onset Infection | Day 1 to Day 28 (or hospital discharge, if earlier)
  May be further sub-grouped by: pancreatic, peripancreatic, and extra-pancreatic infections, as data allow.
Change in Modified Marshall Score | From Baseline through Day 28 (or hospital discharge, if earlier)
Change in Sequential Organ Failure Assessment (SOFA) Score | From Baseline through Day 28 (or hospital discharge, if earlier)
Change in Systemic Inflammatory Response Syndrome (SIRS) Assessment | From Baseline through Day 28 (or hospital discharge, if earlier)
Change in Abdominal Pain Numeric Rating Score | From Baseline through Day 28 (or hospital discharge, if earlier)
Change in Computed Tomography Severity Index (CTSI) Score for Pancreatitis | From Baseline through Day 60 Follow-up
Change in Modified Computed Tomography Severity Index (mCTSI) Score for Pancreatitis | From Baseline through Day 60 Follow-up

CONTACTS AND LOCATIONS:
Locations (14):
- United States (11):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Keck Hospital of USC and LA County Hospital, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida Health, Gainesville, Florida
  - Orlando Health, Orlando, Florida
  - UI Health, University of Illinois Chicago Hospital Health Sciences System, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Medical Center, New York, New York
- India (3):
  - Lisie Hospital, Kochi, Kerala
  - Christian Medical College (CMC) Vellore, Ranipet Campus, Vellore, TamiNadu
  - All India Institute of Medical Sciences, Delhi

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.